CLINICAL TRIAL: NCT05416398
Title: The Effect of Aerobic and High-Intensity Interval Training on Respiratory Function, Exercise Capacity and Secondary Outcomes in Obstructive Sleep Apnea
Brief Title: Effects of High-intensity Interval Training and Aerobic Exercise on Obstructive Sleep Apnea.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Engin Ramazanoglu, Researcher, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/57
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Function Loss; Exercise Capacity; Fatigue; Selective Attention; Physical Parameters
Keywords: Aerobic Exercise; Exercise Tolerance; High Intensity Interval Training; Obstructive Sleep Apnea
MeSH Terms: conditions — Fatigue; Sleep Apnea, Obstructive | interventions — Exercise; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental model
Who Masked: Participant
Masking Description: After the patients were selected from the relevant population with the improbable random sampling method, the patients who accepted to participate in the study and met the inclusion criteria will be assigned to one of the aerobic exercise group, high-intensity interval training training group or control group with the closed-envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): They will only receive standard medical treatment. In addition to the evaluation parameters applied, no additional information and/or exercise will be recommended other than routine clinical treatment and recommendations.
- Aerobic Exercise (Experimental): Aerobic exercise group; 3 days a week, 45-60 minutes will be carried out in the form of walking and jogging on the treadmill. Initially, warm-up exercises (10 minutes) will perform walking at 35-70% of maximum heart rate (HRmax). Then, aerobic exercises, the resistance and duration of which are increased according to the tolerance of the patient on the treadmill for 30-35 minutes, and at 60-70% of the HRmax, attention will be paid to ensure that the fatigue severity perceived by the patients is within the range of 12-14 according to the Modified Borg scale. Afterwards, the exercise program will be terminated with a cooling period (10 minutes) consisting of walking at a light pace.
  Interventions: Other: Aerobic Exercise, High Intensity Interval Training
- High-İntensity İnterval Training (Experimental): The high-intensity interval training (HIIT) group, it will be performed as walking or jogging on the treadmill for 4X4 minutes (16 minutes in total) at ≥ 80% of HRmax, three times a week, with each session lasting a total of 38 minutes. Each training session will begin with a 10-minute warm-up period at 70% of HRmax. Between each 4-minute interval and after the last interval, patients will walk at 70% of HRmax for 3 minutes. Patients will check heart rate and target heart rate to control exercise intensity and will aim to reach their individual target heart rate after 1-1.5 minutes of exercise in each interval. The physical therapist, who oversees all training sessions, will check the patients' target heart rates.
  Interventions: Other: Aerobic Exercise, High Intensity Interval Training

INTERVENTIONS:
Other: Aerobic Exercise, High Intensity Interval Training — Aerobic exercise is a form of exercise done by consuming oxygen in order to give energy to the body. High Intensity Interval Training consists of low-intensity periods of active rest combined with short periods of intense exercise.
  Arms: Aerobic Exercise; High-İntensity İnterval Training

SUMMARY:
Introduction: Obstructive sleep apnea syndrome (OSAS) is a condition characterized by recurrent episodes of partial or complete obstruction of the upper airway (URI) during sleep.

Objective: It was designed to compare the effects of aerobic and high-intensity interval training training on exercise capacity, fatigue, cognitive status, physical and disease-specific parameters in individuals with obstructive sleep apnea syndrome.

Materials and Methods: It was designed as a randomized controlled experimental model. Patients between the ages of 18-55 who were diagnosed with OSAS by polysomnography by a specialist physician, and those with moderate (AHI: 16-30) and severe (AHI> 30) OSAS will be included. After the patients were selected from the relevant population with the improbable random sampling method, the patients who accepted to participate in the study and met the inclusion criteria will be assigned to one of the aerobic exercise group, high-intensity interval training training group or control group with the closed-envelope method. Evaluations will be evaluated for each group before the first session of the exercise program and one day after the last session after they have completed the 8-week exercise program. Evaluation parameters; 6-minute walk test, fatigue severity scale, stroop test, skinfold, tape measure, comprehensive respiratory function test device (MasterScreen™ Body Plethysmography), Turkish version of the functional outcomes of the disease-specific quality of life sleep questionnaire (functional outcomes of sleep questionnaire, FOSQ,tr) The nottingham health profile includes the Epworth sleepiness scale.

Conclusion: The effects of aerobic and high-intensity interval training training will be interpreted by comparing the evaluations before and after treatment and between groups.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a condition characterized by recurrent episodes of partial or complete obstruction of the upper airway (URI) during sleep. It results in recurrent awakenings and episodic oxyhemoglobin desaturations due to decreased ventilation. Clinical manifestations of the disease are snoring, witnessed apnea, suffocation, night sweats, nocturnal arrhythmias, excessive daytime sleepiness, personality changes, morning headache, decreased decision-making ability, forgetfulness, anxiety, depression, cardiovascular diseases, hypertension, myocardial infarction, cardiac It encompasses a wide spectrum of insufficiency, metabolic dysfunction, and cor pulmonale. There are 3 main causes of upper respiratory tract obstruction. These are the tone of the pharyngeal muscles, negative pressure during inspiration and the anatomical structure of the URI. Pharyngeal obstruction plays the most important role. The pharynx can be thought of as a tube devoid of a bony roof, and its opening is determined by the balance between the forces in the closing direction (such as negative intraluminal pressure and externally compressing adipose tissue) and the dilator muscles.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with moderate (AHI:16-30) and severe (AHI>30) OSAS by polysomnography.
* Patients who are inactive according to the International Physical Activity Questionnaire-Short Form
* Patients with symptoms of Obstructive Sleep Apnea Syndrome (snoring, respiratory arrest, and daytime sleepiness).

Exclusion Criteria:

* Conditions that may make exercise dangerous. Patients with angina pectoris, congestive heart failure, cardiomyopathy, coronary artery disease, emphysema, inflammatory and malignant lung disease, pneumothorax.
* Those with chronic obstructive pulmonary disease
* Those who have recently had upper respiratory tract surgery.
* Those with cooperation problems that would prevent the subject from successfully participating and completing the protocol, such as serious neurological, psychological, and medical problems.
* Uncooperative patients.
* Patients who previously received continuous positive airway pressure therapy
* Behavior therapy training.
* Patients already taking an exercise program.
* Patients who cannot exercise due to musculoskeletal disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Tests | 8 week
  Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and ratios will be used in statistical analysis.(FEV1/FVC)
Exercise Capacity | 8 week
  Exercise capacity will be evaluated with a 6-minute walk test. Evaluates the integrated responses of all systems involved during exercise, including the pulmonary and cardiovascular systems, blood, neuromuscular system, and muscle metabolism.

SECONDARY OUTCOMES:
Fatigue | 8 week
  It will be evaluated with the Fatigue Severity Scale. FSS is the most commonly used scale among the one-dimensional scales developed to assess fatigue.
Selective Attention | 8 week
  The Stroop Test will be used to evaluate selective attention.
Disease-Specific quality of life | 8 week
  Disease-Specific quality of life will be evaluated with Functional Outcomes of Sleep Questionnaire, FOSQ,tr).
General Health-Related Quality of Life | 8 week
  Overall health-related quality of life will be assessed with the Nottingham Health Profile.
Daytime Sleepiness | 8 week
  Epworth Sleepiness Scale will be used to measure the general sleepiness of the patients during the day.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Turgut Özal Medical Center, Department of Chest Diseases, Pulmonary Rehabilitation unit, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will not be shared in order to protect the privacy and confidentiality of patient information.

REFERENCES:
- [Background] Quan SF, O'Connor GT, Quan JS, Redline S, Resnick HE, Shahar E, Siscovick D, Sherrill DL. Association of physical activity with sleep-disordered breathing. Sleep Breath. 2007 Sep;11(3):149-57. doi: 10.1007/s11325-006-0095-5. PMID 17221274
- [Result] Azagra-Calero E, Espinar-Escalona E, Barrera-Mora JM, Llamas-Carreras JM, Solano-Reina E. Obstructive sleep apnea syndrome (OSAS). Review of the literature. Med Oral Patol Oral Cir Bucal. 2012 Nov 1;17(6):e925-9. doi: 10.4317/medoral.17706. PMID 22549673
- [Result] Garcia-Ortega A, Manas E, Lopez-Reyes R, Selma MJ, Garcia-Sanchez A, Oscullo G, Jimenez D, Martinez-Garcia MA. Obstructive sleep apnoea and venous thromboembolism: pathophysiological links and clinical implications. Eur Respir J. 2019 Jan 31;53(2):1800893. doi: 10.1183/13993003.00893-2018. Print 2019 Feb. PMID 30385528
- [Result] Jones RL, Nzekwu MM. The effects of body mass index on lung volumes. Chest. 2006 Sep;130(3):827-33. doi: 10.1378/chest.130.3.827. PMID 16963682